CLINICAL TRIAL: NCT03899220
Title: Addressing Internalized Stigma and Shame as Barriers to Engagement in HIV Care Among Men Who Have Sex With Men (MSM) With Substance Use Disorders (Project Matter)
Brief Title: Project Matter: Intervention to Improve HIV Self-care Among Men Who Have Sex With Men (MSM) With Substance Use Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Abigail Batchelder, Ph.D., M.P.H., Assistant Professor and Staff Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019p001118; K23DA043418 (NIH)
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Substance Use Disorders; HIV/AIDS; Homosexuality, Male
MeSH Terms: conditions — Substance-Related Disorders; Acquired Immunodeficiency Syndrome; Homosexuality, Male

STUDY DESIGN:
Intervention Model Description: Pilot Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This intervention includes 5 face-to-face therapy sessions with a trained clinician plus a bidirectional text component that queries mood, substance use, and medication adherence.
  Interventions: Behavioral: Project Matter
- Enhanced Treatment as Usual (E-TAU) (Active Comparator): Enhanced treatment as usual includes a one session behavioral engagement in care intervention as well as substance use treatment counseling.
  Interventions: Behavioral: Project Matter

INTERVENTIONS:
Behavioral: Project Matter — This intervention includes 5 face-to-face therapy sessions with a trained clinician plus a bidirectional text component that queries mood, substance use, and medication adherence. Both the intervention group and the enhanced treatment as usual (E-TAU) involve a one-session behavioral engagement in care intervention as well as substance use treatment counseling.

SUMMARY:
This study will implement a pilot randomized controlled trial (RCT, N=60) to assess the feasibility and acceptability a refined emotion regulation intervention designed to improve engagement in HIV-care among substance using HIV+ MSM sub-optimally engaged in HIV care.

DETAILED DESCRIPTION:
Eligible study participants will be screened and enrolled at Fenway Health (Boston, MA). Participants will be randomized to an enhanced treatment as usual (E-TAU) arm or the intervention arm. All participants (in both the E-TAU and intervention groups) will receive a one-session behavioral engagement in care intervention, substance use treatment referral information, and the opportunity to discuss and problem solve barriers to substance use treatment with an interventionist, informed by motivational interviewing principles. After randomization, participants in the intervention group will attend 5 therapy sessions focused on behavioral strategies for improving HIV self-care, meta-cognitive awareness of emotions and thoughts, and cognitive restructuring. All participants will receive texts queries about antiretroviral therapy (ART) adherence and substance use, and participants in the intervention group will also receive text queries about mood. All participants will be compensated for every research visit and completed text message blocks.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Cisgender male
* Man who has sex with men (MSM)
* Elevated levels of internalized stigma related to HIV, substance use, or homophobia
* Poorly engaged in HIV care
* Able to provide informed consent
* 18 years or older
* English speaking

Exclusion Criteria:

* Women
* Non-cisgender men
* Do not identify as gay, bisexual, or MSM

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender men who have sex with men
Enrollment: 50 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention | change from baseline to 12 weeks after intervention completion
  The summary score of the Client Satisfaction Questionnaire (CSQ-8) (Sum of 8 questions with response options ranging from 1-4).
Feasibility of Intervention | change from baseline to 12 weeks after intervention completion
  Percent of sessions completed (≥70% considered indicative of feasibility) and percent of text messages responded to by participants (≥70% considered indicative of feasibility).

SECONDARY OUTCOMES:
Engagement in HIV Care | change from baseline to 12 weeks after intervention completion
  Summary Score of 6 indicators of HIV treatment engagement: no missed and not rescheduled HIV-related appointments in the past 3 months, no missed and not rescheduled HIV-related lab tests in the past 3 months, maintaining ART prescriptions over the past 3 months, maintaining >=80% ART adherence in the past 30 days, no period of 4 days where ART was stopped in the past 3 months (without guidance from an HIV care provider), and undetectable viral load at the study visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No